CLINICAL TRIAL: NCT04607408
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of the HIV-1 CH505 Transmitted/Founder gp120 Adjuvanted With GLA-SE in Healthy, HIV-exposed Uninfected Infants
Brief Title: Evaluating Safety and Immune Response to the HIV-1 CH505 Transmitted/Founder gp120 Adjuvanted With GLA-SE in Healthy, HIV-exposed Uninfected Infants
Acronym: HVTN 135
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HIV Vaccine Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 135; UM1AI068614 (NIH)
Record Dates: First submitted 2020-10-16; First posted 2020-10-29 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: HIV Infections
Keywords: HIV; Vaccine; Infant
MeSH Terms: conditions — HIV Infections | interventions — glucopyranosyl lipid-A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Part A, Group 1: CH505TF gp120 + GLA-SE (Experimental): Participants received 20 mcg Stable CH505TF gp120 admixed with 2.5 mcg GLA-SE, administered as a 0.25 mL intramuscular (IM) injection into either thigh at Weeks 0, 8, 16, 32, and 54.
  Interventions: Biological: CH505TF gp120; Biological: GLA-SE adjuvant
- Part A, Group 2: Placebo (Placebo Comparator): Participants received Placebo administered as a 0.25 mL IM injection, into either thigh at Weeks 0, 8, 16, 32, and 54.
  Interventions: Biological: Placebo
- Part B, Group 3: CH505TF gp120 + GLA-SE (Experimental): Participants received 20 mcg Stable CH505TF gp120 admixed with 5 mcg GLA-SE, administered as a 0.5 mL IM injection into either thigh at Weeks 0, 8, 16, 32, and 54.
  Interventions: Biological: CH505TF gp120; Biological: GLA-SE adjuvant
- Part B, Group 4: Placebo (Placebo Comparator): Participants received Placebo administered as a 0.5 mL IM injection, into either thigh at Weeks 0, 8, 16, 32, and 54.
  Interventions: Biological: Placebo
- Part C, Group 5: CH505TF gp120 + GLA-SE (Experimental): Participants received 20 mcg Stable CH505TF gp120 admixed with 5 mcg GLA-SE, administered as a 0.5 mL IM injection into either thigh at Weeks 0, 8, 16, 32, and 54.
  Interventions: Biological: CH505TF gp120; Biological: GLA-SE adjuvant
- Part C, Group 6: Placebo (Placebo Comparator): Participants received Placebo administered as a 0.5 mL IM injection, into either thigh at Weeks 0, 8, 16, 32, and 54.
  Interventions: Biological: Placebo
- Part C, Group 7: CH505TF gp120 + GLA-SE (Experimental): Participants received 5 mcg Stable CH505TF gp120 admixed with 5 mcg GLA-SE, administered as a 0.5 mL IM injection into either thigh at Weeks 0, 8, 16, 32, and 54.
  Interventions: Biological: CH505TF gp120; Biological: GLA-SE adjuvant
- Part C, Group 8: Placebo (Placebo Comparator): Participants received Placebo administered as a 0.5 mL IM injection, into either thigh at Weeks 0, 8, 16, 32, and 54.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CH505TF gp120 — HIV-1 CH505 transmitted/founder virus Env gp120 immunogen
  Arms: Part A, Group 1: CH505TF gp120 + GLA-SE; Part B, Group 3: CH505TF gp120 + GLA-SE; Part C, Group 5: CH505TF gp120 + GLA-SE; Part C, Group 7: CH505TF gp120 + GLA-SE
Biological: GLA-SE adjuvant — An oil-in-water stable emulsion (SE) containing the immunological adjuvant Glucopyranosyl Lipid A (GLA)
  Arms: Part A, Group 1: CH505TF gp120 + GLA-SE; Part B, Group 3: CH505TF gp120 + GLA-SE; Part C, Group 5: CH505TF gp120 + GLA-SE; Part C, Group 7: CH505TF gp120 + GLA-SE
Biological: Placebo — Sodium Chloride for Injection, 0.9% USP
  Arms: Part A, Group 2: Placebo; Part B, Group 4: Placebo; Part C, Group 6: Placebo; Part C, Group 8: Placebo

SUMMARY:
This study evaluated the safety and immune response in healthy HIV-exposed and uninfected infants to the protein vaccine, CH505TF gp120, adjuvanted with GLA-SE.

DETAILED DESCRIPTION:
This study evaluated evaluate the safety and immune response in healthy HIV-exposed and uninfected infants to the protein vaccine, CH505TF gp120, adjuvanted with GLA-SE.

This study enrolled 38 mother-infant pairs. To quantify the maternal HIV antibody response, mothers were also enrolled in the study but not received study product. Infants received the CH505TF gp120 protein adjuvanted with GLA-SE at Weeks 0, 8, 16, 32, and 54. The first dose was given within the first five days of life.

The study was conducted in three parts (Parts A, B, and C), and to ensure safety, enrollment proceeded in stages.

Part A (Initial Safety) enrolled first. 5 infants in Part A received a low dose of protein with a low dose of adjuvant and 2 infants received placebo.

After safety review post first vaccination of infants in Part A, Part B enrolled. In Part B (Safety Ramp-Up), 2 infants received a higher dose of protein with a higher dose of adjuvant and 2 infants received placebo.

After safety review post first vaccination of infants in Part B, Part C enrolled. In Part C (Immunogenicity), 5 infants received low dose protein with higher dose of adjuvant, 16 infants received a higher dose of protein with higher dose of adjuvant, and 6 infants received placebo.

There were 14 scheduled clinic visits over 24.5 months. For infants, study visits included some or all of the following: physical examinations, medical history, vaccine injections, HIV testing, and blood, cord blood, and stool collection. For mothers, study visits included some or all of the following: medical history, physical examinations, questionnaires, risk reduction counseling, and blood, breastmilk, and stool collection.

ELIGIBILITY:
Infant Inclusion Criteria:

* Born via Caesarean section to an HIV-1-infected woman who meets all maternal inclusion/exclusion criteria listed below.
* Estimated gestational age at birth is at least 37 weeks.
* Weight at birth is at least 2.5 kg.
* Has initiated antiretroviral prophylaxis consistent with current site-specific standard of care.
* Hemoglobin >14.0 g/dL.
* White Blood Cell Count ≥ 7000 cells/mm3
* Platelets > 100,000 cells/mm3
* Alanine aminotransferase (ALT) <1.25 times upper limit of age adjusted normal.
* Creatinine < 1.1 times upper limit of age adjusted normal.
* Negative HIV-1 nucleic acid test on specimen drawn within 72 hours of birth.
* Written informed consent provided by mother.
* Age is equal to or less than five days.

Infant Exclusion Criteria:

* Any clinically significant congenital anomaly/birth defect.
* Documented or suspected serious medical illness, infection, clinically significant finding from physical examination or immediate life-threatening condition, including requirement for ongoing supplemental oxygen, as judged by the examining clinician.
* Receipt of or anticipated need for blood products, immunoglobulin, or immunosuppressive therapy. This includes infants who require Hepatitis B Immunoglobulin (HBIG) but does not require exclusion of infants who receive Hepatitis B vaccine in the newborn period.
* Receipt of any other investigational product.

Mother Inclusion Criteria:

* Mother's age is at least 18 years, and willing and able to provide written informed consent for her and her infant's participation in this study.
* Mother is in the second or third trimester of singleton pregnancy, as determined by a clinical exam, or sonography and reported menstrual history.
* Mother agrees to donate umbilical cord blood.
* Mother has a planned Caesarian Section at Chris Hani Baragwanath Academic Hospital, Soweto and plans to remain in the area after delivery.
* Mother is determined by the site investigator to be in good overall health at the time of delivery based on medical history, and physical exam.
* Mother has a documented CD4 count > 350 cells/microliter during her pregnancy.
* Mother has a documented SARS-CoV-2 negative PCR test within 2 days before delivery to 5 days after delivery
* Mother has access to the participating HVTN CRS and willingness to be followed for the planned duration of the study.
* Assessment of understanding: Mother demonstrates understanding of this study; completes a questionnaire prior to delivery with verbal demonstration of understanding of all questionnaire items answered incorrectly.
* Mother agrees not to enroll either herself or her infant in another research study for the duration of the trial without prior approval of the HVTN 135 PSRT.
* Mother has confirmed HIV-1 infection documented by medical records at any time during or prior to screening, and confirmed by the HVTN CRS by serology.
* Mother has been on cART for at least sixteen weeks prior to delivery and intends to continue with cART for the duration of breastfeeding.\
* Mother has a viral load of less than 400 copies/mL between two weeks before and 5 days after delivery.

Mother Exclusion Criteria:

* Any WHO Grade IV illness within one year prior to study enrollment as determined by the history and physical examination and review of the medical record (if available). These include HIV wasting syndrome, PJP Pneumonia, Cerebral Toxoplasmosis, extrapulmonary Cryptococcosis, Progressive Multifocal Leukoencephalopathy, any disseminated endemic mycosis (histoplasmosis), candidiasis of the esophagus, trachea, bronchi or lung, disseminated atypical mycobacteria, non-typhoid Salmonella septicemia, extrapulmonary tuberculosis, lymphoma, Kaposi's sarcoma.
* Prior participation in any HIV-1 vaccine or anti-HIV antibody-mediated prevention trial.
* Receipt of any investigational agent during this pregnancy.
* Receipt of blood products, immunoglobulin, or immunomodulating therapy within 45 days prior to delivery of the placenta.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent.
* Any condition that places the newborn at higher risk of early-onset sepsis, such as concern for active maternal infection at delivery as determined by local site investigators (eg, fever).
* Detectable Hepatitis B surface antigen.

Ages: 0 Days to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avy Violari, Study Chair — Perinatal HIV Research Unit, Chris Hani Baragwanath Hospital; Georgia Tomaras, Study Chair — Duke University, HVTN Laboratory
Locations (1):
- Perinatal HIV Research Unit (PHRU), Soweto CRS, Johannesburg, Gauteng, South Africa

REFERENCES:
- [Derived] Violari A, Otwombe K, Hahn W, Chen S, Josipovic D, Baba V, Angelidou A, Smolen KK, Levy O, Mkhize NN, Woodward Davis AS, Martin TM, Haynes BF, Williams WB, Sagawa ZK, Kublin JG, Polakowski L, Brewinski Isaacs M, Yen C, Tomaras G, Corey L, Janes H, Gray GE. Safety and implementation of phase I randomized GLA-SE-adjuvanted CH505TF gp120 HIV vaccine trial in newborns. J Clin Invest. 2025 Apr 3;135(11):e186927. doi: 10.1172/JCI186927. eCollection 2025 Jun 2. PMID 40178906
- [Derived] Violari A, Otwombe K, Hahn W, Chen S, Josipovic D, Baba V, Angelidou A, Smolen KK, Levy O, Mkhize NN, Woodward AS, Martin TM, Haynes B, Williams WB, Sagawa ZK, Kublin J, Polakowski L, Isaacs MB, Yen C, Tomaras G, Corey L, Janes H, Gray G. Safety and implementation of a phase 1 randomized GLA-SE-adjuvanted CH505TF gp120 HIV vaccine trial in newborns. medRxiv [Preprint]. 2024 Oct 17:2024.10.15.24315548. doi: 10.1101/2024.10.15.24315548. PMID 39484284

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled 38 mother-infant pairs. Mothers were also enrolled to assess maternal HIV antibody response but did not receive study product. All mother-infant pairs were assigned to Groups as a unit. The values reported reflect the number of infants, who were the primary participants. Each infant corresponds to one unique mother, so the number of mothers equals the number of infants.
Groups:
- Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54): Placebo (Sodium Chloride, 0.9% USP) administered as a 0.25 mL (Group 2) or 0.5 mL (Groups 4, 6, and 8) IM injection at Weeks 0, 8, 16, 32, and 54
- Part A, Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54): 20 mcg Stable CH505TF gp120 admixed with 2.5 mcg GLA-SE, administered as a 0.25 mL IM injection into either thigh at Weeks 0, 8, 16, 32, and 54
- Part B, Group 3: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54); Part C, Group 5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54): 20 mcg Stable CH505TF gp120 admixed with 5 mcg GLA-SE, administered as a 0.5 mL IM injection into either thigh at Weeks 0, 8, 16, 32, and 54
- Part C, Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54): 5 mcg Stable CH505TF gp120 admixed with 5 mcg GLA-SE, administered as a 0.5 mL IM injection into either thigh at Weeks 0, 8, 16, 32, and 54
Period: Overall Study
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Part A, Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Part B, Group 3: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Started (The values reported reflect the number of infants, who were the primary participants. Each infant corresponds to one unique mother, so the number of mothers equals the number of infants.) | 10 | 5 | 2 | 16 | 5
Completed (The values reported reflect the number of infants, who were the primary participants. Each infant corresponds to one unique mother, so the number of mothers equals the number of infants.) | 10 | 4 | 2 | 14 | 5
Not Completed | 0 | 1 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented separately for mothers and infants. Mothers were enrolled to assess maternal HIV antibody response and did not receive study product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Part A, Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Part B, Group 3: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Total
Number analyzed (Participants) | 10 | 5 | 2 | 16 | 5 | 38
Age, Continuous [Median (Full Range); unit: days] — Age of Infants (Continuous)
  days | 4 [4 to 5] | 4 [2 to 4] | 4.5 [4 to 5] | 4 [2 to 5] | 4 [3 to 5] | 4 [2 to 5]
Age, Continuous [Median (Full Range); unit: years] — Age of Mothers (Continuous)
  years | 31.5 [26 to 39] | 36 [34 to 38] | 36 [35 to 37] | 34.5 [24 to 41] | 33 [25 to 36] | 34 [24 to 41]
Sex: Female, Male [Count of Participants; unit: Participants] — Sex of Infants (Female, Male)
  Participants
    Female | 6 | 1 | 1 | 9 | 1 | 18
    Male | 4 | 4 | 1 | 7 | 4 | 20
Sex: Female, Male [Count of Participants; unit: Participants] — Sex of Mothers (Female, Male)
  Participants
    Female | 10 | 5 | 2 | 16 | 5 | 38
    Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity of Infants
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 10 | 5 | 2 | 16 | 5 | 38
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity of Mothers
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 10 | 5 | 2 | 16 | 5 | 38
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of Infants
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 10 | 5 | 2 | 16 | 5 | 38
    White | 0 | 0 | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of Mothers
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 10 | 5 | 2 | 16 | 5 | 38
    White | 0 | 0 | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Region of Enrollment of Infants
  Participants
    South Africa | 10 | 5 | 2 | 16 | 5 | 38
Region of Enrollment [Count of Participants; unit: Participants] — Region of Enrollment of Mothers
  Participants
    South Africa | 10 | 5 | 2 | 16 | 5 | 38

OUTCOME MEASURES:

1. Primary Outcome: WHO Anthropometric Measure of Weight-for-Age Z-Score
Description: At each study visit, the infant's weight was measured. Using weight and age, a WHO weight-for-age z-score will be calculated using the World Health Organization (WHO) anthropometric calculator tool. Weight-for-age reflects body weight relative to the child's age on a given day. A Z-score of 0 represents the population mean, a Z-score less than -2 indicates an infant who is underweight, -2 to 2 indicates an infant who is normal weight, and above 2 indicates the infant may have a growth problem, but this is better assessed from weight-for-length.
  This Outcome Measure was not collected for Mothers.
Time Frame: Measured at each study visit.
Population: Safety population
Measure: Median (Full Range); unit: Z-scores
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Part A, Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Part B, Group 3: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 10 | 5 | 2 | 16 | 5
Z-scores
  Screening Visit | -0.32 [-1.15 to 1.47] | -0.80 [-1.54 to 0.51] | -1.59 [-2.1 to -1.08] | -0.29 [-1.47 to 0.82] | 0.60 [-1.22 to 0.87]
  Month 0/Prior to Vaccination 1 | -0.54 [-1.9 to 1.39] | -1.16 [-1.51 to 0.45] | -1.36 [-1.72 to -0.99] | -0.47 [-2.41 to 1.46] | 0.06 [-1.25 to 0.74]
  1 Day Post Vaccination 1 | -0.47 [-1.96 to 1.28] | -1.13 [-1.57 to 0.39] | -1.39 [-1.81 to -0.96] | -0.44 [-1.31 to 0.52] | -0.05 [-1.09 to 0.73]
  14 Days Post Vaccination 1 | -0.50 [-2.14 to 1.42] | -0.53 [-1.55 to 0.89] | -1.02 [-1.09 to -0.95] | -0.29 [-1.37 to 0.83] | 0.03 [-0.61 to 0.4]
  Month 2/Prior to Vaccination 2 | -0.25 [-2.06 to 1.44] | 0.15 [-1.8 to 0.98] | -1.27 [-1.34 to -1.2] | -0.34 [-1.47 to 1.3] | 0.07 [-0.54 to 0.55]
  14 Days Post Vaccination 2 | -0.50 [-2.04 to 1.68] | 0.22 [-1.78 to 0.7] | -1.30 [-1.4 to -1.2] | 0.02 [-1.23 to 1.52] | -0.04 [-0.47 to 0.68]
  Month 4/Prior to Vaccination 3 | -0.04 [-2.2 to 1.64] | -0.44 [-1.02 to 0.35] | -1.43 [-1.69 to -1.16] | -0.38 [-1.39 to 1.67] | -0.31 [-3.16 to 1.05]
  14 Days Post Vaccination 3 | 0.11 [-1.49 to 1.78] | -0.56 [-1.34 to 0.37] | -1.41 [-1.43 to -1.39] | -0.39 [-1.56 to 1.69] | 0.24 [-0.33 to 1.1]
  Month 8/Prior to Vaccination 4 | 0.12 [-2.02 to 1.72] | -0.76 [-1.37 to 0.76] | -1.69 [-1.89 to -1.49] | -0.09 [-1.08 to 2.24] | 0.60 [-0.72 to 1.73]
  14 Days Post Vaccination 4 | 0.23 [-1.82 to 1.67] | -0.69 [-1.41 to 0.75] | -1.71 [-1.73 to -1.69] | -0.04 [-1.28 to 2.29] | -0.20 [-0.72 to 1.59]
  Month 12.5/Prior to Vaccination 5 | -0.03 [-1.87 to 1.67] | -0.25 [-1.83 to 0.13] | -1.30 [-1.32 to -1.27] | 0.29 [-1.61 to 2.2] | -0.14 [-0.48 to 1.35]
  14 Days Post Vaccination 5 | -0.18 [-1.74 to 1.6] | -0.39 [-1.9 to 0.12] | -1.20 [-1.2 to -1.2] | 0.52 [-1.49 to 2.29] | 0.14 [-0.43 to 1.87]
  4.5 Months Post Vaccination 5 | -0.27 [-1.87 to 1.48] | -1.17 [-2.38 to 0.21] | -1.28 [-1.37 to -1.18] | -0.11 [-1.24 to 2.01] | 1.08 [-0.33 to 2.53]
  12.5 Months Post Vaccination 5 | -0.05 [-1.83 to 1.32] | -0.70 [-2.06 to -0.37] | -0.08 [-0.89 to 0.74] | 0.14 [-1.03 to 1.64] | 0.24 [-0.48 to 0.97]

2. Primary Outcome: Number (Percentage) of Participants by WHO Anthropometric Measure of Weight-for-Age Z-Score Categories
Description: At each study visit, the infant's weight was measured. Using weight and age, a WHO weight-for-age z-score was calculated using the World Health Organization (WHO) anthropometric calculator tool. Weight-for-age reflects body weight relative to the child's age on a given day. Z-scores less than -2 indicates an infant who is underweight, -2 to 2 indicates an infant who is normal weight, and above 2 indicates the infant may have a growth problem, but this is better assessed from weight-for-length.
Time Frame: Measured at each study visit.
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54): Placebo (Sodium Chloride, 0.9% USP) to be administered as a 0.25 mL (Group 2) or 0.5 mL (Groups 4, 6, and 8) IM injection at Weeks 0, 8, 16, 32, and 54
- Part A, Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54): 20 mcg Stable CH505TF gp120 admixed with 2.5 mcg GLA-SE, to be administered as a 0.25 mL IM injection into either thigh at Weeks 0, 8, 16, 32, and 54
- Part B, Group 3: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54); Part C, Group 5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54): 20 mcg Stable CH505TF gp120 admixed with 5 mcg GLA-SE, to be administered as a 0.5 mL IM injection into either thigh at Weeks 0, 8, 16, 32, and 54
- Part C, Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54): 5 mcg Stable CH505TF gp120 admixed with 5 mcg GLA-SE, to be administered as a 0.5 mL IM injection into either thigh at Weeks 0, 8, 16, 32, and 54
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Part A, Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Part B, Group 3: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 10 | 5 | 2 | 16 | 5
Participants
  <-2 (Screening Visit) | 0 | 0 | 1 | 0 | 0
  -2 to 2 (Screening Visit) | 10 | 5 | 1 | 16 | 5
  >2 (Screening Visit) | 0 | 0 | 0 | 0 | 0
  <-2 (Month 0/Prior to Vaccination 1) | 0 | 0 | 0 | 1 | 0
  -2 to 2 (Month 0/Prior to Vaccination 1) | 10 | 5 | 2 | 15 | 5
  >2 (Month 0/Prior to Vaccination 1) | 0 | 0 | 0 | 0 | 0
  <-2 (1 Day Post Vaccination 1) | 0 | 0 | 0 | 0 | 0
  -2 to 2 (1 Day Post Vaccination 1) | 10 | 5 | 2 | 16 | 5
  >2 (1 Day Post Vaccination 1) | 0 | 0 | 0 | 0 | 0
  <-2 (14 Days Post Vaccination 1) | 1 | 0 | 0 | 0 | 0
  -2 to 2 (14 Days Post Vaccination 1) | 9 | 5 | 2 | 16 | 5
  >2 (14 Days Post Vaccination 1) | 0 | 0 | 0 | 0 | 0
  <-2 (Month 2/Prior to Vaccination 2): number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  <-2 (Month 2/Prior to Vaccination 2) | 1 | 0 | 0 | 0 | 0
  -2 to 2 (Month 2/Prior to Vaccination 2): number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  -2 to 2 (Month 2/Prior to Vaccination 2) | 9 | 5 | 2 | 15 | 5
  >2 (Month 2/Prior to Vaccination 2): number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  >2 (Month 2/Prior to Vaccination 2) | 0 | 0 | 0 | 0 | 0
  <-2 (14 Days Post Vaccination 2): number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  <-2 (14 Days Post Vaccination 2) | 1 | 0 | 0 | 0 | 0
  -2 to 2 (14 Days Post Vaccination 2): number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  -2 to 2 (14 Days Post Vaccination 2) | 9 | 5 | 2 | 15 | 5
  >2 (14 Days Post Vaccination 2): number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  >2 (14 Days Post Vaccination 2) | 0 | 0 | 0 | 0 | 0
  <-2 (Month 4/Prior to Vaccination 3): number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  <-2 (Month 4/Prior to Vaccination 3) | 1 | 0 | 0 | 0 | 1
  -2 to 2 (Month 4/Prior to Vaccination 3): number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  -2 to 2 (Month 4/Prior to Vaccination 3) | 8 | 5 | 2 | 15 | 3
  >2 (Month 4/Prior to Vaccination 3): number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  >2 (Month 4/Prior to Vaccination 3) | 0 | 0 | 0 | 0 | 0
  <-2 (14 Days Post Vaccination 3): number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  <-2 (14 Days Post Vaccination 3) | 0 | 0 | 0 | 0 | 0
  -2 to 2 (14 Days Post Vaccination 3): number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  -2 to 2 (14 Days Post Vaccination 3) | 9 | 5 | 2 | 15 | 4
  >2 (14 Days Post Vaccination 3): number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  >2 (14 Days Post Vaccination 3) | 0 | 0 | 0 | 0 | 0
  <-2 (Month 8/Prior to Vaccination 4): number analyzed (Participants) | 10 | 5 | 2 | 14 | 5
  <-2 (Month 8/Prior to Vaccination 4) | 1 | 0 | 0 | 0 | 0
  -2 to 2 (Month 8/Prior to Vaccination 4): number analyzed (Participants) | 10 | 5 | 2 | 14 | 5
  -2 to 2 (Month 8/Prior to Vaccination 4) | 9 | 5 | 2 | 13 | 5
  >2 (Month 8/Prior to Vaccination 4): number analyzed (Participants) | 10 | 5 | 2 | 14 | 5
  >2 (Month 8/Prior to Vaccination 4) | 0 | 0 | 0 | 1 | 0
  <-2 (14 Days Post Vaccination 4): number analyzed (Participants) | 10 | 5 | 2 | 14 | 5
  <-2 (14 Days Post Vaccination 4) | 0 | 0 | 0 | 0 | 0
  -2 to 2 (14 Days Post Vaccination 4): number analyzed (Participants) | 10 | 5 | 2 | 14 | 5
  -2 to 2 (14 Days Post Vaccination 4) | 10 | 5 | 2 | 13 | 5
  >2 (14 Days Post Vaccination 4): number analyzed (Participants) | 10 | 5 | 2 | 14 | 5
  >2 (14 Days Post Vaccination 4) | 0 | 0 | 0 | 1 | 0
  <-2 (Month 12.5/Prior to Vaccination 5): number analyzed (Participants) | 10 | 5 | 2 | 13 | 5
  <-2 (Month 12.5/Prior to Vaccination 5) | 0 | 0 | 0 | 0 | 0
  -2 to 2 (Month 12.5/Prior to Vaccination 5): number analyzed (Participants) | 10 | 5 | 2 | 13 | 5
  -2 to 2 (Month 12.5/Prior to Vaccination 5) | 10 | 5 | 2 | 12 | 5
  >2 (Month 12.5/Prior to Vaccination 5): number analyzed (Participants) | 10 | 5 | 2 | 13 | 5
  >2 (Month 12.5/Prior to Vaccination 5) | 0 | 0 | 0 | 1 | 0
  <-2 (14 Days Post Vaccination 5): number analyzed (Participants) | 9 | 5 | 1 | 13 | 5
  <-2 (14 Days Post Vaccination 5) | 0 | 0 | 0 | 0 | 0
  -2 to 2 (14 Days Post Vaccination 5): number analyzed (Participants) | 9 | 5 | 1 | 13 | 5
  -2 to 2 (14 Days Post Vaccination 5) | 9 | 5 | 1 | 12 | 5
  >2 (14 Days Post Vaccination 5): number analyzed (Participants) | 9 | 5 | 1 | 13 | 5
  >2 (14 Days Post Vaccination 5) | 0 | 0 | 0 | 1 | 0
  <-2 (4.5 Months Post Vaccination 5): number analyzed (Participants) | 10 | 4 | 2 | 14 | 5
  <-2 (4.5 Months Post Vaccination 5) | 0 | 1 | 0 | 0 | 0
  -2 to 2 (4.5 Months Post Vaccination 5): number analyzed (Participants) | 10 | 4 | 2 | 14 | 5
  -2 to 2 (4.5 Months Post Vaccination 5) | 10 | 3 | 2 | 13 | 4
  >2 (4.5 Months Post Vaccination 5): number analyzed (Participants) | 10 | 4 | 2 | 14 | 5
  >2 (4.5 Months Post Vaccination 5) | 0 | 0 | 0 | 1 | 1
  <-2 (12.5 Months Post Vaccination 5): number analyzed (Participants) | 10 | 3 | 2 | 14 | 5
  <-2 (12.5 Months Post Vaccination 5) | 0 | 1 | 0 | 0 | 0
  -2 to 2 (12.5 Months Post Vaccination 5): number analyzed (Participants) | 10 | 3 | 2 | 14 | 5
  -2 to 2 (12.5 Months Post Vaccination 5) | 10 | 2 | 2 | 14 | 5
  >2 (12.5 Months Post Vaccination 5): number analyzed (Participants) | 10 | 3 | 2 | 14 | 5
  >2 (12.5 Months Post Vaccination 5) | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: WHO Anthropometric Measure of Weight-for-Length Z-Score
Description: At each study visit, the infant's length and weight was measured. Using these measurements, a WHO weight-for-length z-score was calculated using the World Health Organization (WHO) anthropometric calculator tool. Weight-for-length reflects body weight in proportion to attained growth in length. A Z-score of 0 represents the population mean, a Z-score less than -2 indicates an infant who is wasted, -2 to 2 indicates an infant who is normal weight, and above 2 indicates the infant is overweight.
  This Outcome Measure was not collected for Mothers.
Time Frame: Measured at each study visit.
Population: Safety population
Measure: Median (Full Range); unit: Z-scores
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Part A, Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Part B, Group 3: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 10 | 5 | 2 | 16 | 5
Z-scores
  Screening Visit | 0.97 [-1.19 to 2.32] | -0.95 [-1.63 to 1.08] | -2.30 [-2.37 to -2.22] | 0.50 [-4.04 to 2.84] | 0.93 [-2.94 to 1.75]
  Month 0/Prior to Vaccination 1 | 0.20 [-1.51 to 1.57] | -0.44 [-1.63 to 1.08] | -0.68 [-1.47 to 0.11] | 0.02 [-1.27 to 1.73] | 0.44 [-2.37 to 1.56]
  1 Day Post Vaccination 1 | 0.40 [-1.4 to 1.69] | 0.44 [-1.47 to 1.7] | -0.58 [-1.43 to 0.27] | 0.06 [-1.5 to 1.68] | 0.05 [-2.17 to 1.33]
  14 Days Post Vaccination 1 | 0.53 [-1.02 to 2.82] | 0.84 [-1.8 to 1.16] | 0.50 [-0.01 to 1] | 0.74 [-0.79 to 3.1] | 0.47 [0.14 to 1.76]
  Month 2/Prior to Vaccination 2 | 1.07 [0.54 to 3.36] | 2.43 [-0.2 to 4.95] | 0.89 [0.35 to 1.42] | 1.60 [-0.09 to 3.21] | 1.25 [0.62 to 3.71]
  14 Days Post Vaccination 2 | 1.14 [0.04 to 2.2] | 1.11 [-0.33 to 2.85] | 0.88 [0.67 to 1.08] | 1.41 [0.1 to 3.36] | 1.88 [0.57 to 2.65]
  Month 4/Prior to Vaccination 3 | 1.55 [0.1 to 2.17] | 0.91 [0.21 to 1.48] | 0.82 [0.23 to 1.41] | 1.04 [-1.26 to 4.41] | 0.99 [0.21 to 3.85]
  14 Days Post Vaccination 3 | 1.55 [-0.06 to 2.21] | 0.48 [-0.52 to 1.98] | -0.02 [-0.69 to 0.65] | 1.16 [-0.99 to 2.91] | 0.69 [0.27 to 2.15]
  Month 8/Prior to Vaccination 4 | 1.07 [-1.42 to 2.88] | 0.67 [0.56 to 1.83] | -0.49 [-0.82 to -0.16] | 1.01 [-0.96 to 2.71] | 0.96 [0.44 to 2.9]
  14 Days Post Vaccination 4 | 1.11 [-1.13 to 3] | 0.68 [-0.07 to 1.52] | 0.18 [-0.62 to 0.97] | 0.69 [-1.07 to 2.83] | 0.45 [0.3 to 2.6]
  Month 12.5/Prior to Vaccination 5 | 0.96 [-1.27 to 3.25] | 0.91 [-0.1 to 1.72] | -0.04 [-0.52 to 0.44] | 0.79 [-0.56 to 2.79] | 1.39 [-0.59 to 2.72]
  14 Days Post Vaccination 5 | 0.66 [-0.96 to 2.6] | 0.93 [-0.39 to 1.83] | 0.63 [0.63 to 0.63] | 0.65 [-0.45 to 2.93] | 1.71 [-0.41 to 2.58]
  4.5 Months Post Vaccination 5 | 0.68 [-1.27 to 2.44] | 0.08 [-0.59 to 1.29] | -0.36 [-0.58 to -0.13] | 0.89 [-0.4 to 2.25] | 0.79 [-0.61 to 2.69]
  12.5 Months Post Vaccination 5 | 1.06 [-1.26 to 2.24] | 0.72 [0 to 0.83] | 0.59 [0.34 to 0.83] | 1.05 [-0.2 to 2.27] | 1.70 [-0.26 to 3]

4. Primary Outcome: Number (Percentage) of Participants by WHO Anthropometric Measure of Weight-for-Length Z-Score Categories
Description: At each study visit, the infant's length and weight was measured. Using these measurements, a WHO weight-for-length z-score was calculated using the World Health Organization (WHO) anthropometric calculator tool. Weight-for-length reflects body weight in proportion to attained growth in length. Z-scores less than -2 indicates an infant who is wasted, -2 to 2 indicates an infant who is normal weight, and above 2 indicates the infant is overweight.
Time Frame: Measured at each study visit.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Part A, Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Part B, Group 3: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 10 | 5 | 2 | 16 | 5
Participants
  <-2 (Screening Visit): number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  <-2 (Screening Visit) | 0 | 0 | 2 | 1 | 1
  -2 to 2 (Screening Visit): number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  -2 to 2 (Screening Visit) | 8 | 5 | 0 | 12 | 3
  >2 (Screening Visit): number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  >2 (Screening Visit) | 1 | 0 | 0 | 2 | 0
  <-2 (Month 0/Prior to Vaccination 1): number analyzed (Participants) | 10 | 5 | 2 | 15 | 4
  <-2 (Month 0/Prior to Vaccination 1) | 0 | 0 | 0 | 0 | 1
  -2 to 2 (Month 0/Prior to Vaccination 1): number analyzed (Participants) | 10 | 5 | 2 | 15 | 4
  -2 to 2 (Month 0/Prior to Vaccination 1) | 10 | 5 | 2 | 15 | 3
  >2 (Month 0/Prior to Vaccination 1): number analyzed (Participants) | 10 | 5 | 2 | 15 | 4
  >2 (Month 0/Prior to Vaccination 1) | 0 | 0 | 0 | 0 | 0
  <-2 (1 Day Post Vaccination 1): number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  <-2 (1 Day Post Vaccination 1) | 0 | 0 | 0 | 0 | 1
  -2 to 2 (1 Day Post Vaccination 1): number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  -2 to 2 (1 Day Post Vaccination 1) | 10 | 5 | 2 | 15 | 4
  >2 (1 Day Post Vaccination 1): number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  >2 (1 Day Post Vaccination 1) | 0 | 0 | 0 | 0 | 0
  <-2 (14 Days Post Vaccination 1) | 0 | 0 | 0 | 0 | 0
  -2 to 2 (14 Days Post Vaccination 1) | 9 | 5 | 2 | 14 | 5
  >2 (14 Days Post Vaccination 1) | 1 | 0 | 0 | 2 | 0
  <-2 (Month 2/Prior to Vaccination 2): number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  <-2 (Month 2/Prior to Vaccination 2) | 0 | 0 | 0 | 0 | 0
  -2 to 2 (Month 2/Prior to Vaccination 2): number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  -2 to 2 (Month 2/Prior to Vaccination 2) | 8 | 1 | 2 | 10 | 3
  >2 (Month 2/Prior to Vaccination 2): number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  >2 (Month 2/Prior to Vaccination 2) | 2 | 4 | 0 | 5 | 2
  <-2 (14 Days Post Vaccination 2): number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  <-2 (14 Days Post Vaccination 2) | 0 | 0 | 0 | 0 | 0
  -2 to 2 (14 Days Post Vaccination 2): number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  -2 to 2 (14 Days Post Vaccination 2) | 9 | 4 | 2 | 11 | 3
  >2 (14 Days Post Vaccination 2): number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  >2 (14 Days Post Vaccination 2) | 1 | 1 | 0 | 4 | 2
  <-2 (Month 4/Prior to Vaccination 3): number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  <-2 (Month 4/Prior to Vaccination 3) | 0 | 0 | 0 | 0 | 0
  -2 to 2 (Month 4/Prior to Vaccination 3): number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  -2 to 2 (Month 4/Prior to Vaccination 3) | 8 | 5 | 2 | 12 | 3
  >2 (Month 4/Prior to Vaccination 3): number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  >2 (Month 4/Prior to Vaccination 3) | 1 | 0 | 0 | 3 | 1
  <-2 (14 Days Post Vaccination 3): number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  <-2 (14 Days Post Vaccination 3) | 0 | 0 | 0 | 0 | 0
  -2 to 2 (14 Days Post Vaccination 3): number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  -2 to 2 (14 Days Post Vaccination 3) | 7 | 5 | 2 | 13 | 3
  >2 (14 Days Post Vaccination 3): number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  >2 (14 Days Post Vaccination 3) | 2 | 0 | 0 | 2 | 1
  <-2 (Month 8/Prior to Vaccination 4): number analyzed (Participants) | 10 | 5 | 2 | 14 | 5
  <-2 (Month 8/Prior to Vaccination 4) | 0 | 0 | 0 | 0 | 0
  -2 to 2 (Month 8/Prior to Vaccination 4): number analyzed (Participants) | 10 | 5 | 2 | 14 | 5
  -2 to 2 (Month 8/Prior to Vaccination 4) | 8 | 5 | 2 | 12 | 3
  >2 (Month 8/Prior to Vaccination 4): number analyzed (Participants) | 10 | 5 | 2 | 14 | 5
  >2 (Month 8/Prior to Vaccination 4) | 2 | 0 | 0 | 2 | 2
  <-2 (14 Days Post Vaccination 4): number analyzed (Participants) | 10 | 5 | 2 | 14 | 5
  <-2 (14 Days Post Vaccination 4) | 0 | 0 | 0 | 0 | 0
  -2 to 2 (14 Days Post Vaccination 4): number analyzed (Participants) | 10 | 5 | 2 | 14 | 5
  -2 to 2 (14 Days Post Vaccination 4) | 8 | 5 | 2 | 11 | 3
  >2 (14 Days Post Vaccination 4): number analyzed (Participants) | 10 | 5 | 2 | 14 | 5
  >2 (14 Days Post Vaccination 4) | 2 | 0 | 0 | 3 | 2
  <-2 (Month 12.5/Prior to Vaccination 5): number analyzed (Participants) | 10 | 5 | 2 | 13 | 5
  <-2 (Month 12.5/Prior to Vaccination 5) | 0 | 0 | 0 | 0 | 0
  -2 to 2 (Month 12.5/Prior to Vaccination 5): number analyzed (Participants) | 10 | 5 | 2 | 13 | 5
  -2 to 2 (Month 12.5/Prior to Vaccination 5) | 8 | 5 | 2 | 12 | 4
  >2 (Month 12.5/Prior to Vaccination 5): number analyzed (Participants) | 10 | 5 | 2 | 13 | 5
  >2 (Month 12.5/Prior to Vaccination 5) | 2 | 0 | 0 | 1 | 1
  <-2 (14 Days Post Vaccination 5): number analyzed (Participants) | 9 | 5 | 1 | 13 | 5
  <-2 (14 Days Post Vaccination 5) | 0 | 0 | 0 | 0 | 0
  -2 to 2 (14 Days Post Vaccination 5): number analyzed (Participants) | 9 | 5 | 1 | 13 | 5
  -2 to 2 (14 Days Post Vaccination 5) | 7 | 5 | 1 | 12 | 3
  >2 (14 Days Post Vaccination 5): number analyzed (Participants) | 9 | 5 | 1 | 13 | 5
  >2 (14 Days Post Vaccination 5) | 2 | 0 | 0 | 1 | 2
  <-2 (4.5 Months Post Vaccination 5): number analyzed (Participants) | 10 | 4 | 2 | 14 | 5
  <-2 (4.5 Months Post Vaccination 5) | 0 | 0 | 0 | 0 | 0
  -2 to 2 (4.5 Months Post Vaccination 5): number analyzed (Participants) | 10 | 4 | 2 | 14 | 5
  -2 to 2 (4.5 Months Post Vaccination 5) | 9 | 4 | 2 | 11 | 3
  >2 (4.5 Months Post Vaccination 5): number analyzed (Participants) | 10 | 4 | 2 | 14 | 5
  >2 (4.5 Months Post Vaccination 5) | 1 | 0 | 0 | 3 | 2
  <-2 (12.5 Months Post Vaccination 5): number analyzed (Participants) | 10 | 3 | 2 | 14 | 5
  <-2 (12.5 Months Post Vaccination 5) | 0 | 0 | 0 | 0 | 0
  -2 to 2 (12.5 Months Post Vaccination 5): number analyzed (Participants) | 10 | 3 | 2 | 14 | 5
  -2 to 2 (12.5 Months Post Vaccination 5) | 9 | 3 | 2 | 12 | 3
  >2 (12.5 Months Post Vaccination 5): number analyzed (Participants) | 10 | 3 | 2 | 14 | 5
  >2 (12.5 Months Post Vaccination 5) | 1 | 0 | 0 | 2 | 2

5. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The maximum grade observed for each symptom over the time frame is presented.
  This Outcome Measure was not collected for Mothers.
Time Frame: Measured through 7 days after each vaccine dose (Weeks 0, 8, 16, 32, 54).
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Part A, Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Part B, Group 3: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 10 | 5 | 2 | 16 | 5
Participants
  None | 9 | 4 | 2 | 12 | 5
  Mild | 1 | 1 | 0 | 3 | 0
  Moderate | 0 | 0 | 0 | 1 | 0
  Severe | 0 | 0 | 0 | 0 | 0
  Potentially Life-threatening | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 5
Time Frame: Measured through 7 days after each vaccine dose (Weeks 0, 8, 16, 32, 54).
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Part A, Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Part B, Group 3: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 10 | 5 | 2 | 16 | 5
Participants
  Erythema/redness: None | 10 | 3 | 2 | 16 | 5
  Erythema/redness: Mild | 0 | 2 | 0 | 0 | 0
  Erythema/redness: Moderate | 0 | 0 | 0 | 0 | 0
  Erythema/redness: Severe | 0 | 0 | 0 | 0 | 0
  Erythema/redness: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Induration/swelling: None | 10 | 5 | 2 | 16 | 5
  Induration/swelling: Mild | 0 | 0 | 0 | 0 | 0
  Induration/swelling: Moderate | 0 | 0 | 0 | 0 | 0
  Induration/swelling: Severe | 0 | 0 | 0 | 0 | 0
  Induration/swelling: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 10 | 3 | 2 | 16 | 5
  Erythema and/or Induration: Mild | 0 | 2 | 0 | 0 | 0
  Erythema and/or Induration: Moderate | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: Severe | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The following symptoms are considered as systemic reactogenicity if the onset date was within the periods of assessment specified in the protocol: fever, sleepiness/lethargy, rash, vomiting, anorexia, seizure. The item Max. Systemic Symptoms is the maximum of the individual systemic reactogenicities for a participant.
  This Outcome Measure was not collected for Mothers.
Time Frame: Measured through 7 days after each vaccine dose (Weeks 0, 8, 16, 32, 54).
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Part A, Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Part B, Group 3: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 10 | 5 | 2 | 16 | 5
Participants
  Anorexia: None | 9 | 5 | 2 | 11 | 5
  Anorexia: Mild | 1 | 0 | 0 | 5 | 0
  Anorexia: Moderate | 0 | 0 | 0 | 0 | 0
  Anorexia: Severe | 0 | 0 | 0 | 0 | 0
  Anorexia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Fever: None | 8 | 5 | 2 | 15 | 2
  Fever: Mild | 2 | 0 | 0 | 1 | 3
  Fever: Moderate | 0 | 0 | 0 | 0 | 0
  Fever: Severe | 0 | 0 | 0 | 0 | 0
  Fever: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Rash: None | 8 | 5 | 2 | 13 | 5
  Rash: Mild | 2 | 0 | 0 | 3 | 0
  Rash: Moderate | 0 | 0 | 0 | 0 | 0
  Rash: Severe | 0 | 0 | 0 | 0 | 0
  Rash: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Seizure: None | 10 | 5 | 2 | 16 | 5
  Seizure: Mild | 0 | 0 | 0 | 0 | 0
  Seizure: Moderate | 0 | 0 | 0 | 0 | 0
  Seizure: Severe | 0 | 0 | 0 | 0 | 0
  Seizure: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Sleepiness/lethargy: None | 7 | 5 | 2 | 13 | 3
  Sleepiness/lethargy: Mild | 3 | 0 | 0 | 3 | 1
  Sleepiness/lethargy: Moderate | 0 | 0 | 0 | 0 | 1
  Sleepiness/lethargy: Severe | 0 | 0 | 0 | 0 | 0
  Sleepiness/lethargy: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Vomiting: None | 10 | 4 | 2 | 15 | 3
  Vomiting: Mild | 0 | 1 | 0 | 1 | 2
  Vomiting: Moderate | 0 | 0 | 0 | 0 | 0
  Vomiting: Severe | 0 | 0 | 0 | 0 | 0
  Vomiting: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0
  Max. Systemic Sypmtoms: None | 6 | 4 | 2 | 8 | 2
  Max. Systemic Sypmtoms: Mild | 4 | 1 | 0 | 8 | 2
  Max. Systemic Sypmtoms: Moderate | 0 | 0 | 0 | 0 | 1
  Max. Systemic Sypmtoms: Severe | 0 | 0 | 0 | 0 | 0
  Max. Systemic Sypmtoms: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number (Percentage) of Participants With Local Laboratory Values Recorded as Meeting Grade 1 AE Criteria or Above as Specified in the Division of AIDS Table.
Description: The number (percentage) of participants with local laboratory values recorded as meeting Grade 1 AE criteria or above as specified in the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events for alanine aminotransferase (ALT), creatinine, hemoglobin, lymphocyte count, neutrophil count, platelets, white blood cells (WBC) was summarized by treatment arm for each post vaccination time point.
  This Outcome Measure was not collected for Mothers.
Time Frame: ALT, creatinine, hemoglobin, platelets, and WBC measured at Screening (Day 0) and Days 14, 70, 126, 238, 393, 743; Lymphocytes and Neutrophils measured at Days 14, 70, 126, 238, 393, 743.
Population: 'Overall Number of Participants Analyzed' represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, missed the scheduled visit, or terminated participation in the study prior to the scheduled visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Part A, Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Part B, Group 3: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 10 | 5 | 2 | 16 | 5
Participants
  ALT (U/L) - Screening | 0 | 0 | 0 | 0 | 0
  ALT (U/L) - Day 14: number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  ALT (U/L) - Day 14 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) - Day 70: number analyzed (Participants) | 10 | 5 | 2 | 14 | 5
  ALT (U/L) - Day 70 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) - Day 126: number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  ALT (U/L) - Day 126 | 2 | 0 | 0 | 0 | 0
  ALT (U/L) - Day 238: number analyzed (Participants) | 10 | 5 | 2 | 14 | 5
  ALT (U/L) - Day 238 | 1 | 0 | 0 | 0 | 0
  ALT (U/L) - Day 393: number analyzed (Participants) | 9 | 5 | 1 | 13 | 5
  ALT (U/L) - Day 393 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) - Day 743: number analyzed (Participants) | 10 | 3 | 2 | 14 | 5
  ALT (U/L) - Day 743 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) - Screening | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) - Day 14: number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  Creatinine (mg/dL) - Day 14 | 1 | 0 | 0 | 1 | 0
  Creatinine (mg/dL) - Day 70: number analyzed (Participants) | 10 | 5 | 2 | 14 | 5
  Creatinine (mg/dL) - Day 70 | 0 | 0 | 0 | 0 | 1
  Creatinine (mg/dL) - Day 126: number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  Creatinine (mg/dL) - Day 126 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) - Day 238: number analyzed (Participants) | 10 | 5 | 2 | 14 | 5
  Creatinine (mg/dL) - Day 238 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) - Day 393: number analyzed (Participants) | 9 | 5 | 1 | 13 | 5
  Creatinine (mg/dL) - Day 393 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) - Day 743: number analyzed (Participants) | 10 | 3 | 2 | 14 | 5
  Creatinine (mg/dL) - Day 743 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) - Screening | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) - Day 14: number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  Hemoglobin (g/dL) - Day 14 | 7 | 0 | 1 | 7 | 3
  Hemoglobin (g/dL) - Day 70: number analyzed (Participants) | 10 | 4 | 2 | 14 | 5
  Hemoglobin (g/dL) - Day 70 | 4 | 1 | 1 | 7 | 3
  Hemoglobin (g/dL) - Day 126: number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  Hemoglobin (g/dL) - Day 126 | 2 | 0 | 1 | 2 | 0
  Hemoglobin (g/dL) - Day 238: number analyzed (Participants) | 9 | 5 | 1 | 14 | 5
  Hemoglobin (g/dL) - Day 238 | 0 | 1 | 0 | 2 | 0
  Hemoglobin (g/dL) - Day 393: number analyzed (Participants) | 8 | 5 | 1 | 13 | 5
  Hemoglobin (g/dL) - Day 393 | 1 | 0 | 0 | 1 | 0
  Hemoglobin (g/dL) - Day 743: number analyzed (Participants) | 10 | 3 | 2 | 14 | 5
  Hemoglobin (g/dL) - Day 743 | 2 | 1 | 1 | 2 | 0
  Lymphocytes (cells/cubic mm) - Day 14: number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  Lymphocytes (cells/cubic mm) - Day 14 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm) - Day 70: number analyzed (Participants) | 10 | 4 | 2 | 14 | 5
  Lymphocytes (cells/cubic mm) - Day 70 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm) - Day 126: number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  Lymphocytes (cells/cubic mm) - Day 126 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm) - Day 238: number analyzed (Participants) | 9 | 5 | 1 | 14 | 5
  Lymphocytes (cells/cubic mm) - Day 238 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm) - Day 393: number analyzed (Participants) | 8 | 5 | 1 | 13 | 5
  Lymphocytes (cells/cubic mm) - Day 393 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (cells/cubic mm) - Day 743: number analyzed (Participants) | 10 | 3 | 2 | 14 | 5
  Lymphocytes (cells/cubic mm) - Day 743 | 0 | 0 | 0 | 0 | 0
  Neutrophils (cells/cubic mm) - Day 14: number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  Neutrophils (cells/cubic mm) - Day 14 | 0 | 0 | 0 | 1 | 0
  Neutrophils (cells/cubic mm) - Day 70: number analyzed (Participants) | 10 | 4 | 2 | 14 | 5
  Neutrophils (cells/cubic mm) - Day 70 | 1 | 1 | 0 | 0 | 0
  Neutrophils (cells/cubic mm) - Day 126: number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  Neutrophils (cells/cubic mm) - Day 126 | 2 | 2 | 0 | 2 | 0
  Neutrophils (cells/cubic mm) - Day 238: number analyzed (Participants) | 9 | 5 | 1 | 14 | 5
  Neutrophils (cells/cubic mm) - Day 238 | 1 | 0 | 0 | 0 | 0
  Neutrophils (cells/cubic mm) - Day 393: number analyzed (Participants) | 8 | 5 | 1 | 13 | 5
  Neutrophils (cells/cubic mm) - Day 393 | 1 | 0 | 0 | 1 | 0
  Neutrophils (cells/cubic mm) - Day 743: number analyzed (Participants) | 10 | 3 | 2 | 14 | 5
  Neutrophils (cells/cubic mm) - Day 743 | 0 | 0 | 0 | 0 | 0
  Platelets (cells/cubic mm) - Screening | 0 | 0 | 0 | 0 | 0
  Platelets (cells/cubic mm) - Day 14: number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  Platelets (cells/cubic mm) - Day 14 | 0 | 0 | 0 | 0 | 0
  Platelets (cells/cubic mm) - Day 70: number analyzed (Participants) | 10 | 4 | 2 | 14 | 5
  Platelets (cells/cubic mm) - Day 70 | 0 | 0 | 0 | 0 | 0
  Platelets (cells/cubic mm) - Day 126: number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  Platelets (cells/cubic mm) - Day 126 | 0 | 0 | 0 | 1 | 0
  Platelets (cells/cubic mm) - Day 238: number analyzed (Participants) | 9 | 5 | 1 | 14 | 5
  Platelets (cells/cubic mm) - Day 238 | 0 | 0 | 0 | 0 | 0
  Platelets (cells/cubic mm) - Day 393: number analyzed (Participants) | 8 | 5 | 1 | 13 | 5
  Platelets (cells/cubic mm) - Day 393 | 0 | 0 | 0 | 0 | 0
  Platelets (cells/cubic mm) - Day 743: number analyzed (Participants) | 9 | 3 | 2 | 13 | 5
  Platelets (cells/cubic mm) - Day 743 | 0 | 0 | 0 | 0 | 0
  WBC (cells/cubic mm) - Screening | 0 | 0 | 0 | 0 | 0
  WBC (cells/cubic mm) - Day 14: number analyzed (Participants) | 10 | 5 | 2 | 15 | 5
  WBC (cells/cubic mm) - Day 14 | 0 | 0 | 0 | 0 | 0
  WBC (cells/cubic mm) - Day 70: number analyzed (Participants) | 10 | 3 | 2 | 14 | 5
  WBC (cells/cubic mm) - Day 70 | 0 | 0 | 0 | 0 | 0
  WBC (cells/cubic mm) - Day 126: number analyzed (Participants) | 9 | 5 | 2 | 15 | 4
  WBC (cells/cubic mm) - Day 126 | 0 | 0 | 0 | 0 | 0
  WBC (cells/cubic mm) - Day 238: number analyzed (Participants) | 9 | 5 | 1 | 14 | 5
  WBC (cells/cubic mm) - Day 238 | 0 | 0 | 0 | 0 | 0
  WBC (cells/cubic mm) - Day 393: number analyzed (Participants) | 8 | 5 | 1 | 13 | 5
  WBC (cells/cubic mm) - Day 393 | 0 | 0 | 0 | 0 | 0
  WBC (cells/cubic mm) - Day 743: number analyzed (Participants) | 10 | 3 | 2 | 14 | 5
  WBC (cells/cubic mm) - Day 743 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants Reporting AEs, by Highest Severity Grade Per Participant.
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 (exceptions apply).
  This Outcome Measure was not collected for Mothers.
Time Frame: Comprises the entire study period for each infant participant (from the infant's study enrollment until his or her study completion or discontinuation), up to 25 months.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Part A, Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Part B, Group 3: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 10 | 5 | 2 | 16 | 5
Participants
  Mild | 1 | 2 | 0 | 5 | 1
  Moderate | 5 | 2 | 1 | 7 | 4
  Severe | 4 | 1 | 1 | 4 | 0
  Potentially life-threatening | 0 | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0 | 0
  No AE reported | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants Reporting Adverse Events (AEs), by Relationship to Study Product
Description: as for outcome 9
Time Frame: as for outcome 9
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Part A, Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Part B, Group 3: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 10 | 5 | 2 | 16 | 5
Participants
  Related | 1 | 0 | 0 | 0 | 0
  Not Related | 9 | 5 | 2 | 16 | 5
  No AE reported | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: as for outcome 9
Time Frame: as for outcome 9
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Part A, Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Part B, Group 3: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 10 | 5 | 2 | 16 | 5
Participants | 3 | 0 | 1 | 2 | 0

12. Primary Outcome: Magnitude of HIV-1 Env gp120, CD4 Binding Site and V1V2-specific Serum IgG Binding Antibodies, as Assessed by BAMA Two Weeks After the 5th Vaccination
Description: Serum HIV-1-specific IgG responses were measured on a BioPlex instrument (BioRad) using a standardized custom HIV-1 Luminex assay. The readout was background-subtracted mean fluorescence intensity (MFI), where background referred to a plate level control. Net MFI less than 1 is set to 1, and net MFI > 22,000 is set to 22,000. The area under the curve (AUC) was calculated for each participant and antigen using the trapezoidal rule, where the x-axis is log10 dilution and the y-axis is the Net MFI with negative values set to 0. AUC is considered the primary measure of response magnitude.
Time Frame: Measured at month 13, 2 weeks after the 5th vaccination.
Population: "Overall Number of Participants Analyzed" includes those with samples collected at 2 weeks after the 5th vaccination, who were HIV-uninfected and received the last vaccination with specimens. "Number Analyzed" counts participants with available data after filtering for assay-specific quality control criteria. Groups 3 and 5 (20 mcg CH505TF gp120 and 2.5 mcg GLA-SE) who received the same vaccine regimen were pooled in the analyses.
Measure: Median (Inter-Quartile Range); unit: net MFI*log10(dilution)
Groups:
- Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54): 20 mcg Stable CH505TF gp120 admixed with 2.5 mcg GLA-SE, administered as a 0.25 mL IM injection into either thigh at Weeks 0, 8, 16, 32, and 54
- Groups 3+5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54): 20 mcg Stable CH505TF gp120 admixed with 5 mcg GLA-SE, administered as a 0.5 mL IM injection into either thigh at Weeks 0, 8, 16, 32, and 54
- Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54): 5 mcg Stable CH505TF gp120 admixed with 5 mcg GLA-SE, administered as a 0.5 mL IM injection into either thigh at Weeks 0, 8, 16, 32, and 54
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Groups 3+5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 9 | 5 | 14 | 5
net MFI*log10(dilution)
  1086C D7gp120 | 5.2 [3.2 to 8.4] | 16956.7 [16512.5 to 26189.1] | 24059.2 [21832.9 to 30626.7] | 24508.6 [17065.5 to 26209.8]
  CH0505 CON D7gp120 | 3 [1.4 to 6.5] | 7675.3 [6092.5 to 13038.8] | 16065.3 [12036.4 to 24331.6] | 16516.7 [15930.1 to 19086.2]
  CH505TF.6R.SOSIP.664.v4.1 | 19 [2.9 to 221.5] | 50.8 [0.2 to 107.8] | 71.8 [17.4 to 236.6] | 167.8 [93.8 to 188.1]
  Con 6 gp120/B | 7.5 [3.1 to 8.3] | 2333.2 [2327.7 to 2708] | 9386.3 [3803.9 to 15816.8] | 5373.1 [4490.3 to 6747.2]
  Con S gp140 CFI | 7.2 [6.3 to 31] | 8289.3 [2393.4 to 8637.3] | 13322.4 [11569.8 to 23320.6] | 17231.6 [11565.6 to 26860.3]
  gp41 | 2842.4 [2098.3 to 6013.8] | 1670.1 [1031.3 to 2167.9] | 2462 [1603.2 to 3552] | 2251.7 [2095.7 to 2592.4]
  gp70 CH505TF V1V2 | 36.8 [1.9 to 91.3] | 2500.7 [826.8 to 8369.1] | 5768.7 [3342.3 to 9254.4] | 8417 [7400.9 to 22426.2]

13. Primary Outcome: Quantification and Phenotypic Characterization of Peripheral B Cells Capable of Binding HIV-1 Env gp120 and the CD4 Binding Site, as Assessed by Flow Cytometry Two Weeks After the 3rd Vaccination
Description: HIV-1 Env-specific B cells induced by vaccination were identified and characterized using fluorescently labeled recombinant Env proteins in the context of a flow cytometry panel to identify and characterize those B cell. Total B cells are identified using doublet exclusion, lymphocyte scatter profile, a viability dye to exclude dead cells, and are negative for lineage markers: CD3, CD56 and CD14; and positive for CD19 and CD20. B cells are further gated as IgD-, then IgG+, and IgA+.
Time Frame: Measured at month 4.5 (2 weeks post the 3rd vaccination).
Population: "Overall Number of Participants Analyzed" includes those with samples collected at 2 weeks after the 3rd vaccination, who were HIV-uninfected and received the 3rd vaccination with specimens. "Number Analyzed" counts participants with available data after filtering for assay-specific quality control criteria. Groups 3 and 5 (20 mcg CH505TF gp120 and 2.5 mcg GLA-SE) who received the same vaccine regimen were pooled in the analyses.
Measure: Median (Inter-Quartile Range); unit: Percentage of B cells
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Groups 3+5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 9 | 4 | 17 | 4
Percentage of B cells
  CD4-BS specific of B cells | 0.01 [0.01 to 0.01] | 0.02 [0.01 to 0.03] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.02]
  CD4-BS specific of IgA B cells | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0.12]
  CD4-BS specific of IgD- B cells | 0 [0 to 0.01] | 0.25 [0.06 to 0.48] | 0.03 [0.02 to 0.1] | 0.12 [0.03 to 0.36]
  CD4-BS specific of IgG+ B cells | 0 [0 to 0] | 0.71 [0.18 to 1.41] | 0.39 [0.08 to 0.62] | 0.31 [0.06 to 0.77]
  CD4-BS specific of Plasmablasts | 0.05 [0 to 0.06] | 0.03 [0 to 0.07] | 0 [0 to 0.02] | 0 [0 to 0.02]
  CH505+ of B cells | 0.01 [0.01 to 0.01] | 0.09 [0.06 to 0.12] | 0.03 [0.02 to 0.05] | 0.06 [0.05 to 0.08]
  CH505+ of IgA+ B cells | 0 [0 to 0] | 0 [0 to 0.04] | 0 [0 to 0] | 0.18 [0 to 0.51]
  CH505+ of IgD- B cells | 0.01 [0 to 0.01] | 1.98 [1.1 to 2.78] | 0.38 [0.28 to 0.83] | 1.34 [1.1 to 2.1]
  CH505+ of IgG+ B cells | 0 [0 to 0] | 5.98 [3.02 to 8.6] | 3.2 [1.65 to 4.76] | 5.11 [3.29 to 6.6]
  CH505+ of Plasmablasts | 0.06 [0.02 to 0.09] | 0.08 [0.06 to 0.09] | 0.05 [0.02 to 0.07] | 0 [0 to 0.02]
  IgG+ B cells of total B cells | 0.82 [0.61 to 0.87] | 1.41 [1.26 to 1.5] | 0.72 [0.57 to 0.94] | 1.26 [0.95 to 1.49]
  Plasmablasts of B cells | 1.22 [0.54 to 2.13] | 1.24 [1.2 to 1.29] | 0.84 [0.57 to 1.11] | 0.78 [0.45 to 1.21]

14. Primary Outcome: Quantification and Phenotypic Characterization of Peripheral B Cells Capable of Binding HIV-1 Env gp120 and the CD4 Binding Site, as Assessed by Flow Cytometry Two Weeks After the 5th Vaccinations
Description: as for outcome 13
Time Frame: Measured at month 13 (2 weeks after the 5th vaccination).
Population: "Overall Number of Participants Analyzed" includes those with samples collected at 2 weeks after the 5th vaccination, who were HIV-uninfected and received the 5th vaccination with specimens. "Number Analyzed" counts participants with available data after filtering for assay-specific quality control criteria. Groups 3 and 5 (20 mcg CH505TF gp120 and 2.5 mcg GLA-SE) who received the same vaccine regimen were pooled in the analyses.
Measure: Median (Inter-Quartile Range); unit: Percentage of B cells
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Groups 3+5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 9 | 5 | 14 | 5
Percentage of B cells
  CD4-BS specific of B cells | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.02] | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01]
  CD4-BS specific of IgA B cells | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  CD4-BS specific of IgD- B cells | 0 [0 to 0] | 0.06 [0.05 to 0.07] | 0.06 [0.03 to 0.11] | 0.03 [0.03 to 0.04]
  CD4-BS specific of IgG+ B cells | 0 [0 to 0] | 0.12 [0.11 to 0.12] | 0.12 [0.05 to 0.24] | 0.06 [0.04 to 0.07]
  CD4-BS specific of Plasmablasts | 0.04 [0.03 to 0.05] | 0.02 [0 to 0.05] | 0.05 [0.04 to 0.08] | 0.02 [0.01 to 0.13]
  CH505+ of B cells | 0.01 [0.01 to 0.01] | 0.13 [0.05 to 0.23] | 0.07 [0.04 to 0.11] | 0.09 [0.08 to 0.1]
  CH505+ of IgA+ B cells | 0 [0 to 0.04] | 0 [0 to 0] | 0 [0 to 0.06] | 0 [0 to 0.03]
  CH505+ of IgD- B cells | 0 [0 to 0.01] | 0.89 [0.44 to 1.88] | 0.89 [0.49 to 1.15] | 0.8 [0.79 to 0.84]
  CH505+ of IgG+ B cells | 0 [0 to 0] | 2.17 [1.21 to 3.19] | 1.85 [1.32 to 2.78] | 1.7 [1.6 to 1.77]
  CH505+ of Plasmablasts | 0.05 [0.04 to 0.12] | 0.09 [0.05 to 0.12] | 0.12 [0.08 to 0.16] | 0.13 [0.08 to 0.19]
  IgG+ B cells of total B cells | 3.24 [2.87 to 3.75] | 4.42 [4.21 to 6.47] | 3.18 [2.1 to 4.07] | 4.05 [3.7 to 5.27]
  Plasmablasts of B cells | 1.94 [1.3 to 2.37] | 1.87 [1.86 to 1.89] | 1.88 [1.49 to 2.27] | 1.47 [1.33 to 2.06]

15. Secondary Outcome: EPI Vaccine-specific Antibody Responses, as Assessed by Pediatric Vaccine Multiplex Assay (PVMA) 2 Weeks After the 5th Vaccination (Diptheria, HepB, Pertussis, Rubella, and Tetanus)
Description: PVMA uses the same Luminex instrument and techniques as HVTN's standard Binding Antibody Multiplex Assay (BAMA) to assess serum samples for antibodies against diphtheria, tetanus, pertussis, and rubella. The assay is a reliable, high-throughput technique that requires minimal sample volume and measures multiple antibody concentrations. A Hepatitis B antigen was tested as part of the PVMA panel, but did not pass lab-internal QC. The lab opted to test this antigen via ELISA and reported those calculated concentration data for analysis in lieu of the HepB PVMA data. A HepB standard was used in each assay for quality control.
Time Frame: Measured at month 13, 2 weeks after the 5th vaccination.
Population: "Overall Number of Participants Analyzed" includes those with samples collected at 2 weeks after the 5th vaccination, who were HIV-uninfected and received the last vaccination with specimens. "Number Analyzed" counts participants who received all relevant recommended EPI vaccine doses prior to month 13 for a given antigen. Groups 3 and 5 (20 mcg CH505TF gp120 and 2.5 mcg GLA-SE) who received the same vaccine regimen were pooled in the analyses.
Measure: Median (Inter-Quartile Range); unit: IU/mL
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Groups 3+5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 9 | 5 | 14 | 5
IU/mL
  Diptheria: number analyzed (Participants) | 8 | 5 | 13 | 5
  Diptheria | 0.5 [0.4 to 1] | 0.5 [0.4 to 0.9] | 0.3 [0.3 to 0.5] | 0.8 [0.4 to 0.9]
  HepB: number analyzed (Participants) | 8 | 5 | 13 | 5
  HepB | 0.7 [0.4 to 1.1] | 0.1 [0.1 to 0.7] | 0.6 [0.1 to 1] | 0.1 [0.1 to 0.5]
  Pertussis: number analyzed (Participants) | 8 | 5 | 13 | 5
  Pertussis | 5.4 [3.8 to 6.3] | 4.7 [4.1 to 6.2] | 5.8 [3.7 to 7.4] | 7.5 [7.4 to 18.4]
  Rubella | 2.2 [1.3 to 3.2] | 1.4 [0.6 to 1.5] | 1.2 [0.6 to 2.1] | 1.4 [0.6 to 1.6]
  Tetanus: number analyzed (Participants) | 8 | 5 | 13 | 5
  Tetanus | 0.2 [0.1 to 0.3] | 0.3 [0.1 to 0.4] | 0.2 [0.1 to 0.3] | 0.2 [0.1 to 0.2]

16. Secondary Outcome: EPI Vaccine-specific Antibody Responses, as Assessed by Pediatric Vaccine Multiplex Assay (PVMA) 2 Weeks After the 5th Vaccination (HiB and RSV)
Description: PVMA uses the same Luminex instrument and techniques as HVTN's standard Binding Antibody Multiplex Assay (BAMA) to assess serum samples for antibodies against Haemophilus influenzae type B (HiB) and respiratory syncytial virus (RSV). The assay is a reliable, high-throughput technique that requires minimal sample volume and measures multiple antibody concentrations.
Time Frame: Measured at month 13, 2 weeks after the 5th vaccination.
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: µg/mL
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Groups 3+5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 9 | 5 | 14 | 5
µg/mL
  HiB: number analyzed (Participants) | 8 | 5 | 13 | 5
  HiB | 0.2 [0.1 to 0.4] | 0.3 [0 to 0.8] | 0.1 [0 to 0.3] | 0 [0 to 0]
  RSV | 0.2 [0 to 6.2] | 0.4 [0.1 to 4.7] | 4.9 [0.7 to 6.2] | 2.7 [1.7 to 4.4]

17. Secondary Outcome: Magnitude and Breadth of Serum Neutralization of Vaccine-matched Viral Isolates, and Viruses Engineered to Detect Precursors of CD4 Binding Site and V1V2 Antibodies 2 Weeks After the 5th Vaccination.
Description: Neutralizing antibodies against tier 1 and tier 2 strains of HIV-1 were measured as a function of reductions in Tat-regulated luciferase (Luc) reporter gene expression in TZM-bl cells. All serum samples were assayed against Tier 1 and Tier 2 strains of virus by starting with a 1:10 dilution of serum to obtain a neutralizing antibody titer. ID50 (ID80) titers are defined as the serum dilution that reduces RLUs by 50% (or 80%) relative to the RLUs in virus control wells after subtraction of background.
Time Frame: Measured at month 13, 2 weeks after the 5th vaccination.
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: Titers
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Groups 3+5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 9 | 5 | 14 | 5
Titers
  CH0505TF.gly4/GnT1- ID50 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  CH0505TF.gly4/GnT1- ID80 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  CH0505s.G458Y.N279K.2/GnT1 ID50: number analyzed (Participants) | 8 | 5 | 14 | 5
  CH0505s.G458Y.N279K.2/GnT1 ID50 | 11.9 [5 to 19.8] | 5 [5 to 31.7] | 35.4 [19.7 to 64.1] | 28.8 [26 to 36.5]
  CH0505s.G458Y.N279K.2/GnT1 ID80: number analyzed (Participants) | 8 | 5 | 14 | 5
  CH0505s.G458Y.N279K.2/GnT1 ID80 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  CH0505s.G458Y.N279K.N280D.6/GnT1 ID50: number analyzed (Participants) | 5 | 2 | 13 | 5
  CH0505s.G458Y.N279K.N280D.6/GnT1 ID50 | 17.5 [15.4 to 30.6] | 49.1 [34.1 to 64.2] | 32.3 [24 to 56.7] | 29 [25.3 to 31]
  CH0505s.G458Y.N279K.N280D.6/GnT1 ID80: number analyzed (Participants) | 0 | 1 | 3 | 0
  CH0505s.G458Y.N279K.N280D.6/GnT1 ID80 |  | 24 [24 to 24] | 12.9 [12.5 to 15.6] |
  CH505.w4.3 ID50 | 5 [5 to 5] | 481.7 [132.8 to 710.6] | 3961.6 [1226 to 8180.1] | 1157 [681.1 to 2971.8]
  CH505.w4.3 ID80 | 5 [5 to 5] | 86 [22.9 to 115] | 733.9 [214.2 to 1523.5] | 349.7 [93.7 to 445.8]
  CH505TF ID50 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  CH505TF ID80 | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 5]
  CH505TF.gly4.S365P/GnT1- ID50: number analyzed (Participants) | 0 | 1 | 2 | 0
  CH505TF.gly4.S365P/GnT1- ID50 |  | 13.1 [13.1 to 13.1] | 38.8 [34.3 to 43.4] |
  CH505TF.gly4.S365P/GnT1- ID80: number analyzed (Participants) | 0 | 0 | 1 | 0
  CH505TF.gly4.S365P/GnT1- ID80 |  |  | 16.1 [16.1 to 16.1] |

18. Secondary Outcome: Response Rate of Vaccine-elicited Serum Binding Antibodies to FcR Proteins, as Assessed by BAMA 2 Weeks After the 5th Vaccination
Description: Serum HIV-1-specific FcR responses (1:50 dilution) were measured using the standardized custom HIV-1 Luminex assay on a Luminex FLEXMAP 3D system. Readouts were background-subtracted mean fluorescence intensity (MFI), with background defined by plate-level controls. Net MFI was calculated as experimental minus reference antigen MFI, and values <1 were set to 1. Post-enrollment samples were considered positive if they met all three criteria: (1) Net MFI ≥ antigen-specific cutoff (95th percentile of HVTN 115 Part A baseline at Day 0) and ≥ 100 above blank; (2) Net MFI > 3 times the median baseline Net MFI; and (3) MFI > 3 times the median baseline MFI. Response calls were based on the 1:50 dilution. Data were excluded if the blood draw was outside the allowable window, the participant was HIV positive, reference antigen MFI > 5,000, or baseline net MFI > 6,500.
Time Frame: Measured at month 13, 2 weeks after the 5th vaccination.
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Groups 3+5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 9 | 5 | 14 | 5
Participants
  FcGRIIIa F158 1086C D7gp120 | 0 | 5 | 14 | 5
  FcGRIIIa F158 CH0505 CON D7gp120 | 0 | 4 | 14 | 5
  FcGRIIIa F158 CH505TF.6R.SOSIP.664.v4.1 | 0 | 0 | 0 | 0
  FcGRIIIa F158 Con 6 gp120/B | 0 | 0 | 8 | 2
  FcGRIIIa F158 Con S gp140 CFI | 0 | 3 | 14 | 4
  FcGRIIIa F158 gp41 | 3 | 0 | 4 | 1
  FcGRIIIa F158 gp70 CH505TF V1V2 | 0 | 3 | 13 | 5
  FcgRIIa H131 1086C D7gp120 | 0 | 5 | 14 | 5
  FcgRIIa H131 CH0505 CON D7gp120 | 0 | 5 | 14 | 5
  FcgRIIa H131 CH505TF.6R.SOSIP.664.v4.1 | 1 | 1 | 2 | 0
  FcgRIIa H131 Con 6 gp120/B | 0 | 5 | 12 | 5
  FcgRIIa H131 Con S gp140 CFI | 0 | 4 | 14 | 5
  FcgRIIa H131 gp41 | 7 | 2 | 9 | 3
  FcgRIIa H131 gp70 CH505TF V1V2 | 0 | 3 | 13 | 5

19. Secondary Outcome: Magnitude of Vaccine-elicited Serum Binding Antibodies to FcR Proteins, as Assessed by BAMA 2 Weeks After the 5th Vaccination
Description: Serum HIV-1-specific FcR (dilution 1:50) responses were measured on a Luminex FLEXMAP 3D Instrument System using a standardized custom HIV-1 Luminex assay. The readout was background-subtracted mean fluorescence intensity (MFI), where background referred to a plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI less than 1 is set to 1. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI, or baseline net MFI > 6,500.
Time Frame: Measured at month 13, 2 weeks after the 5th vaccination.
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Groups 3+5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 9 | 5 | 14 | 5
relative fluorescence units
  FcGRIIIa F158 1086C D7gp120 | 1 [1 to 1] | 3258.5 [929.5 to 5954.8] | 6725.4 [5105.7 to 10016.2] | 8750.2 [5556.5 to 10306.2]
  FcGRIIIa F158 CH0505 CON D7gp120 | 1 [1 to 1] | 859.2 [157.2 to 1342.2] | 1539.4 [673.2 to 6839.2] | 1922 [1291 to 4116]
  FcGRIIIa F158 CH505TF.6R.SOSIP.664.v4.1 | 1 [1 to 7.5] | 8.8 [7.5 to 11] | 1.6 [1 to 3.8] | 3.8 [1 to 5.3]
  FcGRIIIa F158 Con 6 gp120/B | 1 [1 to 1] | 15.5 [15.3 to 55.5] | 326.1 [31.5 to 3721.7] | 59 [47.8 to 788.2]
  FcGRIIIa F158 Con S gp140 CFI | 1 [1 to 1] | 204 [1 to 512.2] | 422.2 [265.4 to 2271.2] | 1692.8 [445 to 5837.5]
  FcGRIIIa F158 gp41 | 94.8 [47 to 138.2] | 22.5 [17.2 to 26.5] | 45.8 [27.5 to 104.8] | 49.2 [48 to 55]
  FcGRIIIa F158 gp70 CH505TF V1V2 | 1 [1 to 7] | 1323.8 [111.2 to 9646] | 2486.1 [1038.8 to 8161.1] | 6085.2 [4409.8 to 28614.2]
  FcgRIIa H131 1086C D7gp120 | 1 [1 to 1] | 15724.8 [10368.5 to 26417.2] | 27590.1 [24425.3 to 33806.8] | 27235.2 [23596.2 to 33032.5]
  FcgRIIa H131 CH0505 CON D7gp120 | 1 [1 to 1] | 5262 [1516.8 to 9341.8] | 12016.9 [5570.3 to 25277] | 11767.5 [10037 to 16316.2]
  FcgRIIa H131 CH505TF.6R.SOSIP.664.v4.1 | 3 [1 to 33.8] | 18.8 [1 to 34.2] | 9.1 [4.3 to 28.6] | 14.8 [1 to 29]
  FcgRIIa H131 Con 6 gp120/B | 1 [1 to 4.5] | 377.5 [273 to 647.2] | 4278.2 [522.8 to 13886.9] | 860.5 [644.5 to 5295.8]
  FcgRIIa H131 Con S gp140 CFI | 1 [1 to 4] | 4364.5 [227.5 to 5668.5] | 7722.6 [4547.6 to 19637.6] | 12558 [7184 to 25031]
  FcgRIIa H131 gp41 | 306 [125.5 to 693.8] | 94 [65 to 104.5] | 236.6 [64.8 to 565.2] | 338.2 [48 to 383.5]
  FcgRIIa H131 gp70 CH505TF V1V2 | 1 [1 to 2.5] | 5403.8 [311.2 to 22245.2] | 10442.4 [4374.9 to 22312.4] | 16390.8 [15740.5 to 44073.5]

20. Secondary Outcome: Response Rate of Serum Antibody-dependent Cellular Cytotoxicity (ADCC) to CH505TF D7gp120.Avi/293F, as Assessed by Flow Cytometry Assay 2 Weeks After the 5th Vaccination
Description: The qualified GranToxiLux Antibody-Dependent Cell-Mediated Cytotoxicity (ADCC-GTL) assay was performed to measure ADCC-mediated antibody responses. ADCC is quantified as net percent granzyme B activity, which is the percent of target cells positive for GTL (an indicator of granzyme B uptake) minus the percent of target cells positive for GTL when incubated with effector cells in the absence of a source of antibodies. Flow cytometry is used to quantify the frequency of granzyme B positive cells. There is no baseline subtraction applied to the responses, and a fixed positivity threshold is applied to %GzB activity. A positive response is defined as ≥ 8% GzB activity.
Time Frame: Measured at month 13, 2 weeks after the 5th vaccination.
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Groups 3+5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 9 | 5 | 14 | 5
Participants | 0 | 5 | 7 | 0

21. Secondary Outcome: Magnitude of Serum Antibody-dependent Cellular Cytotoxicity (ADCC) to CH505TF D7gp120.Avi/293F, as Assessed by Flow Cytometry Assay 2 Weeks After the 5th Vaccination
Description: The qualified GranToxiLux Antibody-Dependent Cell-Mediated Cytotoxicity (ADCC-GTL) assay was performed to measure ADCC-mediated antibody responses. ADCC is quantified as net percent granzyme B activity, which is the percent of target cells positive for GTL (an indicator of granzyme B uptake) minus the percent of target cells positive for GTL when incubated with effector cells in the absence of a source of antibodies. Flow cytometry is used to quantify the frequency of granzyme B positive cells.
Time Frame: Measured at month 13, 2 weeks after the 5th vaccination.
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: Peak Net % Granzyme B Activity
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Groups 3+5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 9 | 5 | 14 | 5
Peak Net % Granzyme B Activity | 0 [0 to 0.7] | 24.3 [21.8 to 24.5] | 8.1 [5.8 to 9.7] | 6.8 [4.5 to 7]

22. Secondary Outcome: Response Rate of Serum Antibody-dependent Cellular Cytotoxicity (ADCC) to HIV CH0505s.LucR.T2A.Ecto/293T/17, as Assessed by Luciferase Assay 2 Weeks After the 5th Vaccination
Description: ADCC-mediated antibody responses were measured by luciferase ADCC assay using HIV CH0505s.LucR.T2A.ecto/293T/17 Infectious Molecular Clone (IMC)-infected target cells. Luminescence intensity reflects the number of intact target cells remaining after incubation with effector cells in the presence or absence of ADCC-mediating serum antibodies. Lower luminescence corresponds to fewer intact target cells. The outcome measure was calculated as the percent specific change in luciferase activity, defined as: percent specific change in luciferase activity = 100 * (RLU of target and effector well- RLU of test well)/(RLU of target and effector well). There is no baseline subtraction applied to the responses, and a fixed positivity threshold is applied to percent killing or loss of luciferase activity. A positive response is defined as percent specific killing ≥ 15%.
Time Frame: Measured at month 13, 2 weeks after the 5th vaccination.
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Groups 3+5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 9 | 5 | 14 | 5
Participants | 2 | 0 | 4 | 3

23. Secondary Outcome: Magnitude of Serum Antibody-dependent Cellular Cytotoxicity (ADCC) to HIV CH0505s.LucR.T2A.Ecto/293T/17, as Assessed by Luciferase Assay 2 Weeks After the 5th Vaccination
Description: ADCC-mediated antibody responses were measured by luciferase ADCC assay using HIV CH0505s.LucR.T2A.ecto/293T/17 Infectious Molecular Clone (IMC)-infected target cells. Luminescence intensity reflects the number of intact target cells remaining after incubation with effector cells in the presence or absence of ADCC-mediating serum antibodies. Lower luminescence corresponds to fewer intact target cells. The outcome measure was calculated as the percent specific change in luciferase activity, defined as: percent specific change in luciferase activity = 100 * (RLU of target and effector well- RLU of test well)/(RLU of target and effector well).
Time Frame: Measured at month 13, 2 weeks after the 5th vaccination.
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: Peak % loss luciferase activity
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Groups 3+5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 9 | 5 | 14 | 5
Peak % loss luciferase activity | 7.9 [4.9 to 9] | 9 [7.1 to 12.6] | 13.6 [9.5 to 19.9] | 18.4 [14 to 24.7]

24. Secondary Outcome: Response Rate of Serum Antibody-dependent Cellular Phagocytosis (ADCP) to CH505TF D7gp120.Avi/293F, as Assessed by Flow Cytometry 2 Weeks After the 5th Vaccination
Description: ADCP assay is a qualified assay employing flow cytrometric-based technology that measures the ability of antibodies to mediate phagocytosis. A phagocytic score is determined based on the ratio of experimental sample to PBS control. Mean phagocytosis score is defined as: (% bead positive for participant x MFI bead positive for participant) / (% bead positive for PBS only control x MFI bead positive for PBS only control). Higher phagocytosis score values indicate a greater level of antibody-mediated phagocytic activity relative to the PBS control, while values closer to 1 indicate minimal activity above background. Positivity calls were based on two criteria: 1) Average ADCP score ≥ antigen specific cutoff values (max(95th percentile of HVTN 115 baseline ADCP score, 1)) and 2) Average ADCP score > 3x antigen specific median HVTN 115 baseline average ADCP score.
Time Frame: Measured at month 13, 2 weeks after the 5th vaccination.
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Groups 3+5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 9 | 5 | 14 | 5
Participants | 7 | 5 | 14 | 5

25. Secondary Outcome: Magnitude of Serum Antibody-dependent Cellular Phagocytosis (ADCP) to CH505TF D7gp120.Avi/293F, as Assessed by Flow Cytometry 2 Weeks After the 5th Vaccination
Description: ADCP assay is a qualified assay employing flow cytrometric-based technology that measures the ability of antibodies to mediate phagocytosis. A phagocytic score is determined based on the ratio of experimental sample to PBS control. Mean phagocytosis score is defined as: (% bead positive for participant x MFI bead positive for participant) / (% bead positive for PBS only control x MFI bead positive for PBS only control). Higher phagocytosis score values indicate a greater level of antibody-mediated phagocytic activity relative to the PBS control, while values closer to 1 indicate minimal activity above background.
Time Frame: Measured at month 13, 2 weeks after the 5th vaccination.
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: Mean phagocytosis score
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Groups 3+5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
Number analyzed (Participants) | 9 | 5 | 14 | 5
Mean phagocytosis score | 2.1 [1.5 to 2.5] | 14.7 [4.3 to 16.6] | 11.4 [9.1 to 13.9] | 10.9 [10.5 to 11.6]

ADVERSE EVENTS:
Time Frame: The AE reporting period for this study comprises the entire study period for each infant participant (from the infant's study enrollment until his or her study completion or discontinuation), up to 25 months. Reactogenicity events (solicited AEs) were collected through 7 full days after each vaccination. Adverse Event was not collected for Mothers.
Arm/Group | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) | Part A, Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) | Part B, Group 3: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) | Part C, Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5 | 0/2 | 0/16 | 0/5
Serious Adverse Events (participants affected / at risk) | 3/10 | 0/5 | 1/2 | 2/16 | 0/5
Other Adverse Events (participants affected / at risk) | 10/10 | 5/5 | 2/2 | 16/16 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) (N=10) | Part A, Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) (N=5) | Part B, Group 3: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) (N=2) | Part C, Group 5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) (N=16) | Part C, Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) (N=5)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ophthalmia neonatorum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Groups 2, 4, 6, 8: Placebo at w(0,8,16,32,54) (N=10) | Part A, Group 1: 20 mcg CH505TF gp120, 2.5 mcg GLA-SE at w(0,8,16,32,54) (N=5) | Part B, Group 3: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) (N=2) | Part C, Group 5: 20 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) (N=16) | Part C, Group 7: 5 mcg CH505TF gp120, 5 mcg GLA-SE at w(0,8,16,32,54) (N=5)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (10) | 2 (3) | 0 (0) | 2 (2) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post-tussive vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Teething (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Solicited) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site erythema (Solicited) (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (Solicited) (General disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (Solicited) (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus hepatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (4) | 1 (3) | 1 (1) | 3 (3) | 2 (3)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 1 (3) | 1 (1) | 4 (5) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (2) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 6 (11) | 4 (8) | 2 (4) | 4 (10) | 3 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 9 (16) | 3 (4) | 2 (4) | 12 (18) | 4 (5)
Neutrophil count decreased (Investigations) | 6 (6) | 2 (3) | 1 (1) | 4 (7) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Solicited) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Underweight (Metabolism and nutrition disorders) | 4 (7) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Somnolence (Solicited) (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2) | 0 (0) | 2 (3) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3) | 1 (2) | 3 (3) | 1 (1)
Rash (Solicited) (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT04607408/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT04607408/SAP_001.pdf